CLINICAL TRIAL: NCT07345611
Title: Efficacy and Safety of Entecavir With or Without Pegylated Interferon α-2b in Children Aged 3 to 6 Years With Chronic Hepatitis B in the Immune-Clearance Phase (B-Young-Cure-2): A Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Entecavir With or Without Pegylated Interferon α-2b in Children Aged 3-6 Years With Immune-Active Chronic Hepatitis B
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qing-Lei Zeng (Other)
Collaborators: Henan Provincial People's Hospital (Other); Luoyang Central Hospital (Other); Xuchang Central Hospital (Unknown); Luohe Central Hospital (Unknown); Yongcheng People's Hospital (Unknown); Sanmenxia Central Hospital (Unknown); The Third Affiliated Hospital of Henan Medical University (Unknown); Weishi County People's Hospital (Unknown); The Sixth People's Hospital of Zhengzhou (Other); The First Affiliated Hospital of Henan Medical University (Unknown); Shangcheng County People's Hospital (Unknown); The First Affiliated Hospital of Henan Polytechnic University (Unknown); Nanyang Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Qing-Lei Zeng, Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-1631-001
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B Virus Infection; Children; Chronic Hepatitis B
Keywords: Children; Efficacy; Immune clearance; Safety; Chronic; Entecavir; Pegylated interferon α-2b; Functional cure; Hepatitis B virus
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic; Bronchiolitis Obliterans Syndrome | interventions — entecavir

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir (Experimental): Receive entecavir monotherapy throughout the 96-week treatment course.
  Interventions: Drug: Entecavir
- Entecavir plus Peg-IFN α-2b (Experimental): Receive entecavir for the first 48 weeks, followed by combination therapy with pegylated interferon α-2b for the remaining 48 weeks.
  Interventions: Drug: Entecavir + Pegylated interferon α-2b

INTERVENTIONS:
Drug: Entecavir — Receive entecavir onotherapy throughout the 96-week treatment course, the dosage of entecavir is 0.015 mg/kg/day for those weighing between 10 and 30 kg; for those weighing more than 30 kg, the dosage is 0.5 mg/day, oral.
  Other Names: Runzhong®
  Arms: Entecavir
Drug: Entecavir + Pegylated interferon α-2b — Receive entecavir (with dosing adjusted by body weight: 0.015 mg/kg/day for subjects weighing 10-30 kg, and 0.5 mg/day for those >30 kg, oral) for the first 48 weeks, followed by combination therapy with pegylated interferon α-2b (104 μg/m², weekly, subcutaneous injection) for the remaining 48 weeks.
  Other Names: Runzhong®; PEGBING®
  Arms: Entecavir plus Peg-IFN α-2b

SUMMARY:
This study aims to evaluate the efficacy and safety of entecavir monotherapy versus sequential entecavir plus pegylated interferon α-2b in achieving functional cure in immune-active, HBeAg-positive children aged 3-6 years with chronic hepatitis B.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized controlled, phase 4 trial enrolling 3-6-year-old children with HBeAg-positive CHB in the immune-clearance phase. Participants will be randomly assigned in a 1:1 ratio to two treatment arms, both lasting 96 weeks. The ETV group will receive entecavir (ETV) monotherapy throughout the 96-week treatment course (ETV group). The pegylated interferon (Peg-IFN) group will receive ETV for the first 48 weeks, followed by combination therapy with Peg-IFN α-2b for the remaining 48 weeks (ETV plus IFN combination group). The primary endpoint is the functional cure rate at 24 weeks after treatment discontinuation (week 120). The main secondary endpoints include the rates of undetectable HBV DNA, HBeAg loss, and HBsAg loss at week 24, 48, 72, 96, and 120, and rates of alanine aminotransferase elevation or flares (>5 times of upper limit of normal) and incidence of adverse events at any time during the study. The study will also explore associations between functional cure and baseline or on-treatment parameters. A total of 80 children (40 per group) is required to detect a statistically significant difference between two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 and 6 (more than 3 but less than 7) years;
2. Chronic HBV infection;
3. Positive HBeAg;
4. HBV DNA >1.0×10⁴ IU/mL;
5. Normal upper abdominal ultrasound without cirrhosis or hepatocellular carcinoma;
6. ALT >40 U/L.

Exclusion Criteria:

1. Previous antiviral treatment for chronic HBV infection;
2. Coinfection with hepatitis C, D, E, human immunodeficiency virus (HIV), Epstein-Barr virus, or cytomegalovirus;
3. Previous or current evidence of hepatocellular carcinoma or cirrhosis;
4. Coexistence of any other liver diseases such as autoimmune hepatitis, drug-induced liver injury or Wilson's disease;
5. Coexistence of systemic/other organ disorders (for example with evidence of thyroid disorders);
6. Hemoglobin level <100 g/L;
7. Absolute neutrophil count <1.0×10⁹/L.;
8. Platelet count <125×10⁹/L;
9. Total bilirubin >1 ULN, i.e., 17.1 μmol/L;
10. Albumin level <35 g/L;
11. Concurrent treatment with other drugs, including but not limited to nephrotoxic drugs, immune modulators, cytotoxic drugs, Chinese traditional medicine or supplements, nonsteroidal anti-inflammatory drugs, or steroids.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-11 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of functional cure | At 24 weeks after treatment cessation.
  Functional cure is defined as the loss of HBsAg to <0.05 IU/mL and HBeAg clearance, with or without the presence of hepatitis B surface antibody (HBsAb) and hepatitis B e antibody (HBeAb), and undetectable HBV DNA (<10 IU/mL) at the end of treatment, sustained through 24 weeks post-treatment.

SECONDARY OUTCOMES:
The rate of HBV DNA undetectable | At week 24, 48, 72, 96, 120 of the study.
  Proportion of participants with HBV DNA undetectable, defined as HBV DNA <10 IU/mL.
The rate of HBeAg loss | At week 24, 48, 72, 96, 120 of the study.
  Proportion of participants with HBeAg loss, defined as HBeAg <0.18 PEIU/mL.
The rate of HBsAg loss | At week 24, 48, 72, 96, 120 of the study.
  Proportion of participants with HBsAg loss, defined as HBsAg <0.05 IU/mL.
The rate of alanine aminotransferase elevation or flare | At any time during the study, i.e., from the date of patient enrollment through 24 weeks after treatment discontinuation.
  Proportion of participants with alanine aminotransferase elevation (> 1 time the upper limit of normal, i.e., >40 U/L) or flare rate, defined as ALT >5 times the upper limit of normal (ULN), i.e., >200 U/L.
The rate of cytopenia rate | At any time during the study, i.e., from the date of patient enrollment through 24 weeks after treatment discontinuation.
  Proportion of participants with cytopenia, defined as an absolute neutrophil count <1.0×10⁹/L and/or a platelet count <100×10⁹/L.
The rate of growth suppression | At week 24, 48, 60, 72, 84, 96, 108, 120 of the study.
  Growth suppression rate, defined as height and weight measurements falling below expected levels based on Chinese national standards and World Health Organization anthropometric z-scores for child growth.
The rate of thyroid dysfunction | At week 72, 96, and 120 of the study.
  Proportion of participants with thyroid dysfunction rate, defined as thyroid-stimulating hormone (TSH, normal range 0.27-10 mU/L), free thyroxine (FT4, normal range 10.3-31 pmol/L), or free triiodothyronine (FT3, normal range 3-11.4 pmol/L) levels exceeds the limit of normal or the lower limit of normal .
Any other adverse event | At any time during study, i.e., from the date of patient enrollment through 24 weeks after treatment discontinuation.
  Incidence of other adverse event at any time during study, including but not limited to flu-like symptoms and signs, rash, and other expected or unexpected adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Qing-Lei Zeng, M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No